CLINICAL TRIAL: NCT04864769
Title: Effect of Intake of Hydrolyzed Krill Protein Isolate, Whey Protein Isolate and Soy Protein Isolate on Plasma Amino Acid Profile
Brief Title: Effect of Intake of Hydrolyzed Krill Protein Isolate on Plasma Amino Acid Profile
Acronym: KRILL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mette Hansen (Other)
Collaborators: Aker BioMarine Human Ingredients AS (Industry)
Responsible Party: Sponsor-Investigator, Mette Hansen, Associate Professor, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Krill Protein
Record Dates: First submitted 2021-04-13; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Human Nutrition
Keywords: Protein; Amino Acids; Krill; Whey; Soy; Satiety; Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Soybean Proteins; Water

STUDY DESIGN:
Intervention Model Description: Design and Method: Randomized, controlled, double-blind cross-study, in which 12 healthy adult young men in randomized order ingest 35 g of protein of crude protein from one of the three protein sources or water on four different experimental days. Before and up to three hours after ingestion of the test beverage, blood samples are collected for 8 time points during each experimental day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Krill Protein Hydrolysate (Experimental): Krill Protein Hydrolysate
  Interventions: Dietary Supplement: Krill protein hydrolysate
- Soy protein isolate (Active Comparator): Soy Protein isolate
  Interventions: Dietary Supplement: Soy protein isolate
- Whey protein isolate (Active Comparator): Whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate
- Control (Sham Comparator): Water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Krill protein hydrolysate — Ingestion of 35 g Krill protein hydrolysate
  Arms: Krill Protein Hydrolysate
Dietary Supplement: Soy protein isolate — Ingestion of 35 g Soy protein isolate
  Arms: Soy protein isolate
Dietary Supplement: Whey protein isolate — Ingestion of 35 g Whey protein isolate
  Arms: Whey protein isolate
Dietary Supplement: Water — Ingestion of water (control)
  Arms: Control

SUMMARY:
Purpose: To examine the absorption of three different protein sources: hydrolyzed krill protein isolate, whey protein isolate, and soy protein isolate.

DETAILED DESCRIPTION:
Design and Method: Randomized, controlled, double-blind cross-study, in which 12 healthy adult young men in randomized order ingest 35 g of protein of crude protein from one of the three protein sources or water on four different experimental days. Before and up to three hours after ingestion of the test beverage, blood samples are collected for 8 time points during each experimental day.

ELIGIBILITY:
Inclusion Criteria:

* men
* 18-30 years

Exclusion Criteria:

* smoking,
* medication,
* health issues conflicting with the experimental trial

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Amino acids concentrations | 10 minutes prior to supplement up to 180 minutes after supplement
  Measurement of changes in amino acids concentrations in the blood

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 10 minutes prior to supplement up to 180 minutes after supplement
  Measurements of changes in Hunger and satiety using 100 mm Visual Analogue Scores
Insulin | 10 minutes prior to supplement up to 180 minutes after supplement
  Changes in serum insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available by contacting the corresponding author up to five years after publication. However, before reuse an acceptance from the participants for reuse is mandatory.